CLINICAL TRIAL: NCT04080284
Title: Trial of Maintenance With Niraparib in Patients With Stage III, Stage IV or Platinum-sensitive Recurrent Uterine Serous Carcinoma
Brief Title: Trial of Maintenance With Niraparib- Uterine Serous Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Principal Investigator, Marina Frimer, Principle Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0380
Record Dates: First submitted 2019-08-15; First posted 2019-09-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer; Papillary Serous Endometrial Carcinoma; Uterine Serous Carcinoma; Endometrial Carcinoma; Cancer of the Endometrium
Keywords: Niraparib; uterine Cancer; papillary serous uterine cancer; endometrial cancer; serous uterine cancer; Endometrial; Endometrial Carcinoma; Recurrent Uterine Carcinoma; platinum-sensitive
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: Niraparib maintenance treatment will be given to patients for 1 year on study or until disease progression. Patients not tolerating the treatment will stop the niraparib treatment based on criteria described below. Patients who are benefitting from treatment will have access to their assigned treatment as long as considered acceptable by their treating physician or until they are discontinued for one of the below reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Niraparib (Experimental): Oral niraparib
  -Cohort - Uterine serous carcinoma
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Study treatment will be administered orally Q day continuously. Up to three capsules of 100mg strength will be taken at each dose administration. Initiation dose will be defined per current FDA guidelines for Niraparib treatment in ovarian cancer. Dose interruption (no longer than 28 days) will be allowed. Dose reduction will be allowed based on treatment side effects. Dose reductions to 2 capsules daily (200mg) and subsequently to 1 capsule daily (100mg) will be allowed. No further dose reductions will be allowed. The timing of efficacy or safety evaluations should not be affected by dose interruptions or reductions.
  Other Names: ZEJULA

SUMMARY:
Uterine serous carcinoma (USC) accounts for up to 40% of endometrial cancer-related deaths. Patients with USC share many genomic and clinical characteristics with patients who has serous ovarian cancer. The objective of this study is to evaluate the efficacy of maintenance Niraparib regimen in patients with advanced or platinum sensitive recurrent uterine serous carcinoma. Additionally, the investigators aim to further describe the safety of this regimen. The investigators hypothesize that Niraparib maintenance will be a well-tolerated treatment and show significant response in patients with uterine serous carcinoma.

DETAILED DESCRIPTION:
Uterine serous carcinoma (USC) accounts for up to 40% of endometrial cancer-related deaths. In contrast to the more common endometrioid histology, USC is more likely to present in advanced stage and carries a worse prognosis. USC mimics the most common serous carcinoma of the ovary and has high probability for nodal and intra-peritoneal spread. Furthermore, studies have indicated that USC harbors a high frequency of somatic TP53 mutations, germline BRCA1 mutations, and mutations within the Fanconi Anemia - BRCA pathway. Data is supportive of the USC association with hereditary breast and ovarian cancer, essentially harboring mutations in DNA repair genes. Approximately 5% of women with USC have germline mutations in 3 different tumor suppressor genes including BRCA1, CHEK2, and TP53.(1,2) The Cancer Genome Atlas Research network reported 4 groups of endometrial tumors based on integrated genomic data - including a novel POLE subtype in 10% endometrial tumors. Patients with uterine serous cancers shared many similar characteristics with basal-like breast and high grade serous ovarian cancers, suggesting a correlation with "BRCAness".(3)

Given the "BRCAness" of USC, recent multicenter prospective cohort study of 1083 women with BRCA1 and BRCA2 mutations who underwent risk reducing salpingo-oophorectomies (RRSO) without hysterectomy were noted to have increased serous/serous-like endometrial carcinoma if they harbored BRCA1 mutations.(4) The study recommended to consider this risk of uterine cancer when discussing the advantages and risks of hysterectomy at the time of RRSO in BRCA1 women. This further supports the high rates of mutations noted among USC patients. A recent systematic review and meta-analysis support the view that USC is a component of BRCA 1/2 -associated tumors. Furthermore, this analysis supports that women with USC should be offered screening for germline mutations when there is a positive family history of malignancies associated with hereditary breast and ovarian cancer syndrome(HBOCS).(5) Furthermore, the Cancer Genome Atlas Research network reported 4 groups of endometrial tumors based on integrated genomic data - including a novel POLE subtype in 10% endometrial tumors. Patients with uterine serous cancers shared many similar characteristics with basal-like breast and high grade serous ovarian cancers, suggesting a correlation with "BRCAness".(3)

Poly(ADP-ribose) polymerases (PARP1 and PARP2) play an important role in DNA repair. Upon formation of DNA breaks, PARP binds at the end of broken DNA strands helping in DNA repair of damage. The hypothesis is that treatment with PARP inhibitors will allow the killing of a subset of cancer cells with deficiencies in DNA repair pathways. For example, a tumor harboring a BRCA or Homologous Recombination gene mutation will have selective blockage by PARP inhibitors in order to maintain genomic integrity. Furthermore, the data in serous ovarian cancer has indicated that tumors arising in a non-BRCA patient that has a homologous recombination deficiency could also enhance tumor cell sensitivity to PARP inhibitors.

PARP inhibitors (PARPi) are synthetically lethal to tumor cells with homologous recombination deficiency (HRD). HRD leads to common phenotype of genome-wide loss of heterozygosity (LOH). Recent analysis of the ARIEL2 part 1 in platinum sensitive ovarian cancer trial found that patients with germline or somatic BRCA mutation or wild-type BRCA with high LOH had longer progression-free survival and improved responses with rucaparib treatment than did patients with wild-type BRCA and low LOH.(7)

The rationale for this current trial is based on significant clinical and genomic similarities of USC and epithelial ovarian carcinomas.(1,2,4) Currently the treatment for stage III and IV USC yields approximately 20-30% survival at 2 years and 10%-20% survival at 3-5 years post diagnosis with current standard therapy of chemotherapy +/-radiation depending on the sites of the disease at surgical staging/debulking. Furthermore, there is no successful second line therapy for patients with recurrent USC and no available clinical trials for patients with recurrent disease. Given the most recent findings of the multi-national, Phase 3 NOVA trial in women with platinum sensitive, recurrent ovarian cancer, Niraparib significantly prolonged the median progression-free survival - irrespective of the presence or absence of a germline BRCA mutation or the presence/absence of a homologous recombinant deficiency.(6) The investigators hypothesize that patients receiving Niraparib maintenance in addition to standard therapy for USC may lead to improved progression free survival in women with suboptimally debulked stage III, stage IV, and platinum-sensitive recurrent USC. The investigators hypothesize that this treatment will be well tolerated in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age at least 18 years
2. ECOG performance status of <2
3. Written voluntary informed consent
4. Histologically diagnosed Uterine Serous Carcinoma.
5. Patient must agree to undergo Foundation One testing.
6. Patient diagnosed with advanced stage USC including stage III, stage IV, or platinum-sensitive recurrent USC
7. If recurrent USC, patient must have platinum sensitive disease after initial treatment; defined as achieving a response (CR or PR) and disease progression >6 months after completion of their last dose of platinum chemotherapy.
8. Patients eligible if receiving 1st or 2nd line chemotherapy for recurrence.
9. The patient must have achieved a partial, stable, or complete tumor response following the last chemotherapy (minimal of 3 cycles) regimen of physician choice chemotherapy indicating partial, stable, complete tumor response.
10. Patients must receive Niraparib maintenance within 12 weeks after completion of their final dose of chemotherapy regimen or within 14 weeks if received radiation therapy. CT Chest/Abd/Pelvis will be performed within 28 days of starting Niraparib.
11. Lesions can be non-measurable or measurable by RECIST 1.1 criteria.
12. Adequate organ function, defined as:

    1. Absolute neutrophil count ≥ 1,500/μL
    2. Platelets ≥ 100,000/μL
    3. Hemoglobin ≥ 9 g/dL
    4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
    5. Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
    6. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
13. Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
14. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
15. Female participant has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non childbearing potential. Non childbearing potential is defined as follows (by other than medical reasons):

    1. ≥45 years of age and has not had menses for >1 year Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See Section 6.4 for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
    2. Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
    3. Able to take oral medications.

Exclusion Criteria:

* 1. Participant must not be simultaneously enrolled in any interventional clinical trial

  2. Drainage of ascites during the last 2 cycles of last chemotherapy

  3. Radiotherapy was given within 2 weeks encompassing >20% of the bone marrow or any radiation therapy within one week prior to Day 1 of protocol therapy. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy.

  4. Persistent >Grade 2 anemia, neutropenia, or thrombocytopenia from prior cancer therapy, that has persisted > 4 weeks and was related to the most recent treatment.

  5. Symptomatic uncontrolled brain or leptomeningeal metastases.

  6. Known hypersensitivity to the components of Niraparib

  7. Major surgery within 3 weeks of starting the study or patient has not recovered from any effects of any major surgery

  8. Diagnosis, detection, or treatment of invasive cancer other than uterine cancer </= 2 years prior to study enrollment (except basal or squamous cell carcinoma of the skin that has been definitively treated)

  9. Patient considered a poor medical risk due to serious, uncontrolled medical disorder, non-malignant systemic disease or active uncontrolled infection.

  10. Patients must not have received a transfusion within 4 weeks of the first dose of study treatment

  11. Participant must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.

  12. Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)

  13. Immunocompromised patients (splenectomy patients are allowed)

  14. Patients with known active hepatitis disease

  15. Prior treatment with a known PARP inhibitor

  16. Patients noted to have MSI-H mutational burden.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
PFS | 1 year
  To determine the Progression Free Survival (PFS) at 1 year in the proposed Niraparib regimen in the population of patients with stage III, all stage IV, or recurrent uterine serous carcinoma (USC).

SECONDARY OUTCOMES:
PFS | 3 years
  Progression-free survival (PFS)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  To further describe safety and assess toxicities encountered with the use of the proposed treatment regimen in patients with stage III, all stage IV, or recurrent uterine serous carcinoma (USC).
Mutational burden | 3 years
  To identify the prevalence of somatic mutations, HRD mutations, and overall mutational burden in patients with USC and classify tumor into loss of heterozygosity (LOH) high and low phenotype.
Quality of Life (QOL) measures using Functional Assessment of Cancer Therapy (FACT- endometrial cancer) and EQ-5D-5L Euroqol | 5 years
  To evaluate quality of life (QOL) for the subjects undergoing this treatment, using validated tools. QOL will be assessed every 3 months during treatment course. [Functional Assessment of Cancer Therapy - Endometrial Cancer questionnaire (score range from 0 to 120 - Higher scores represent better quality of life. EQ-5D-5L Euroqol is scored 0-20, with negative values corresponding to death, full health, and health states worse than death
Overall Survival | 3 years
  Overall Survival
ORR | 3 years
  Overall response rate (ORR) at 2, and 3 years interval from start of treatment protocol

CONTACTS AND LOCATIONS:
Overall Officials: Marina Frimer, MD, Principal Investigator — Northwell Health
Locations (6):
- United States (6):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers NJ School of Medicine, Newark, New Jersey
  - Imbert Cancer Center Northwell Health, Bay Shore, New York
  - Greenlawn Cancer Institute, Northwell Health, Greenlawn, New York
  - RJ Zuckerberg Cancer Hospital, New Hyde Park, New York
  - Cancer Institute at Lenox Hill, New York, New York

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will be available to other researchers via REDCAP, with de-identified source documents uploaded by the site. Remote review of the CRFs will be done monthly, cross-checking with source documents. Clarification of administrative matters will be performed by study coordinator and research manager. Remote monitoring of specific data will include eligibility, adverse events, tumor response, and protocol compliance.
  Data will be maintained in a password- protected secure database, secured on an ePHI. The database will contain a study identifier that is linked to the subject's medical record number. To maintain confidentiality of identifiable information, paper based records will be kept in a secured location only available to research personnel, computer based files will be made available to research personnel through the use of access privileges and passwords, and whenever feasible identifiers will be removed from study information.

REFERENCES:
- [Background] Pennington KP, Walsh T, Lee M, Pennil C, Novetsky AP, Agnew KJ, Thornton A, Garcia R, Mutch D, King MC, Goodfellow P, Swisher EM. BRCA1, TP53, and CHEK2 germline mutations in uterine serous carcinoma. Cancer. 2013 Jan 15;119(2):332-8. doi: 10.1002/cncr.27720. Epub 2012 Jul 18. PMID 22811390
- [Background] Frimer M, Levano KS, Rodriguez-Gabin A, Wang Y, Goldberg GL, Horwitz SB, Hou JY. Germline mutations of the DNA repair pathways in uterine serous carcinoma. Gynecol Oncol. 2016 Apr;141(1):101-7. doi: 10.1016/j.ygyno.2015.12.034. PMID 27016235
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Background] Shu CA, Pike MC, Jotwani AR, Friebel TM, Soslow RA, Levine DA, Nathanson KL, Konner JA, Arnold AG, Bogomolniy F, Dao F, Olvera N, Bancroft EK, Goldfrank DJ, Stadler ZK, Robson ME, Brown CL, Leitao MM Jr, Abu-Rustum NR, Aghajanian CA, Blum JL, Neuhausen SL, Garber JE, Daly MB, Isaacs C, Eeles RA, Ganz PA, Barakat RR, Offit K, Domchek SM, Rebbeck TR, Kauff ND. Uterine Cancer After Risk-Reducing Salpingo-oophorectomy Without Hysterectomy in Women With BRCA Mutations. JAMA Oncol. 2016 Nov 1;2(11):1434-1440. doi: 10.1001/jamaoncol.2016.1820. PMID 27367496
- [Background] de Jonge MM, Mooyaart AL, Vreeswijk MP, de Kroon CD, van Wezel T, van Asperen CJ, Smit VT, Dekkers OM, Bosse T. Linking uterine serous carcinoma to BRCA1/2-associated cancer syndrome: A meta-analysis and case report. Eur J Cancer. 2017 Feb;72:215-225. doi: 10.1016/j.ejca.2016.11.028. Epub 2016 Dec 31. PMID 28049106
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Background] Swisher EM, Lin KK, Oza AM, Scott CL, Giordano H, Sun J, Konecny GE, Coleman RL, Tinker AV, O'Malley DM, Kristeleit RS, Ma L, Bell-McGuinn KM, Brenton JD, Cragun JM, Oaknin A, Ray-Coquard I, Harrell MI, Mann E, Kaufmann SH, Floquet A, Leary A, Harding TC, Goble S, Maloney L, Isaacson J, Allen AR, Rolfe L, Yelensky R, Raponi M, McNeish IA. Rucaparib in relapsed, platinum-sensitive high-grade ovarian carcinoma (ARIEL2 Part 1): an international, multicentre, open-label, phase 2 trial. Lancet Oncol. 2017 Jan;18(1):75-87. doi: 10.1016/S1470-2045(16)30559-9. Epub 2016 Nov 29. PMID 27908594
- [Derived] Takeuchi H, Miyamoto T, Fuseya C, Asaka R, Ida K, Ono M, Tanaka Y, Shinagawa M, Ando H, Asaka S, Shiozawa T. PIM1 is a Poor Prognostic Factor for and Potential Therapeutic Target in Serous Carcinoma of the Endometrium. Int J Gynecol Pathol. 2023 May 1;42(3):282-292. doi: 10.1097/PGP.0000000000000882. Epub 2022 Apr 12. PMID 35443252